CLINICAL TRIAL: NCT04073368
Title: A 16-Week, Single-Blind Randomized, Placebo- Controlled Food Study of the Safety and Tolerability of AXA1125 and AXA1957 in Subjects With Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Study of the Safety and Tolerability of AXA1125 and AXA1957 in Subjects With Non-Alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axcella Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AXA1125-003
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — leucine, isoleucine, valine, arginine, glutamine, and N-acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AXA1957 high dose (Active Comparator): AXA1957 20.3g
  Interventions: Dietary Supplement: AXA1957
- AXA1957 low dose (Active Comparator): AXA1957 13.5g
  Interventions: Dietary Supplement: AXA1957
- AXA1125 (Active Comparator): AXA1125 24g
  Interventions: Dietary Supplement: AXA1125
- Placebo (Placebo Comparator): Placebo 24g
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AXA1957 — Amino acids, food study
  Arms: AXA1957 high dose; AXA1957 low dose
Dietary Supplement: AXA1125 — Amino acids, food study
  Arms: AXA1125
Dietary Supplement: Placebo — Amino acids, food study
  Arms: Placebo

SUMMARY:
This is a randomized, single blind study to determine whether AXA1125 or AXA1957, novel compositions of amino acids, are safe and well tolerated. Subjects have non-alcoholic fatty liver disease (NAFLD) and the study will also examine liver biology using blood tests and magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
This was a 16-week, single-blind, randomized, placebo-controlled food study of the safety and tolerability of AXA1125 and AXA1957 in subjects with NAFLD.

Subjects signed an informed consent form and were screened for eligibility, per the inclusion and exclusion criteria below, up to 6 weeks before the start of the administration period. Subjects were randomized as soon as eligibility was confirmed.

Eligible subjects were randomized in a 2:2:2:1 ratio to receive either AXA1125 24 g twice daily (BID), AXA1957 20.3 g BID, AXA1957 13.5 g BID, or placebo 24 g BID. Randomization occurred via an interactive web response system after eligibility was confirmed and approximately 3 to 5 days prior to the Day 1 visit. Assigned study food product (AXA1125, AXA1957, or placebo) were shipped to the study site upon randomization of each subject.

Once randomization had occurred, subjects presented to the study site on Day 1 (Baseline/Visit 2) for their baseline assessments per the schedule of events. Study Day 1 was the beginning of the 16-week administration period.

Subjects returned to the study site at Week 1 (Visit 3), Week 2 (Visit 4), Week 4 (Visit 5), Week 8 (Visit 6), Week 12 (Visit 7), and Week 16 (Visit 8) to receive their study food product and/or to return any unused study food product, provide blood samples for biomarker and other laboratory testing, undergo liver imaging, and complete other study safety assessments per the schedule of events.

The Safety Follow-up Visit, which occurred approximately 2 weeks after the last visit in the administration period (ie, after the Week 16 visit or at the time of early termination), was the End of Study Visit (Visit 9).

There were 9 study visits in total, including the Screening and Follow-up Visits.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing to participate in the study and provide written informed consent.
* Male and female adults aged > 18 years.
* Subjects must not have participated in any diet/lifestyle intervention or observational studies, or engaged in any body weight altering regimens that resulted in body weight fluctuations (i.e. body weight loss or gain by 5%) in the preceding 3 months prior to Screening.
* A screening MRI consistent with liver inflammation and fibrosis.

Key Exclusion Criteria:

* Current or history of significant alcohol consumption.
* History or presence of liver disease (other than NAFLD/NASH).
* History or presence of cirrhosis and/or history or presence of hepatic decompensation.
* Any diabetes other than Type 2.
* Other poorly controlled medical condition (for example, uncontrolled hypertension with a systolic blood pressure > 100 mmHg).
* Known sensitivity and/or history of clinically significant food intolerance/allergies to proteins (including whey, soy, casein, amino acids, etc.).
* Unable or unwilling to adhere to contraception requirements.
* Any contraindications to a MRI scan.
* Any other condition that, in the opinion of the Investigator, renders the subject at risk for compliance, compromises the well-being of the subject, or hinders study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Harrison, MD, Principal Investigator — Pinnacle Clinical Research
Locations (18):
- United States (18):
  - The Institute for Liver Health LLC, Chandler, Arizona
  - The Institute for Liver Health LLC, Tucson, Arizona
  - National Research Institute, Huntington Park, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - National Research Institute - Panorama, Panorama City, California
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Florida Digestive Health Specialists, Lakewood Rch, Florida
  - Compass Research, LLC - Orlando, Orlando, Florida
  - Bioclinica Research, Orlando, Florida
  - Southern Therapy and Advanced Research LLC, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Gastro One, Germantown, Tennessee
  - Pinnacle Clinical Research, Austin, Texas
  - Liver Center of Texas, Dallas, Texas
  - Doctors Hospital at Renaissance, LLC, Edinburg, Texas
  - Texas Digestive Disease Consultants (TDDC) - Downtown Fort Worth, Fort Worth, Texas
  - Pinnacle Clinical Research, San Antonio, Texas

REFERENCES:
- [Derived] Harrison SA, Baum SJ, Gunn NT, Younes ZH, Kohli A, Patil R, Koziel MJ, Chera H, Zhao J, Chakravarthy MV. Safety, Tolerability, and Biologic Activity of AXA1125 and AXA1957 in Subjects With Nonalcoholic Fatty Liver Disease. Am J Gastroenterol. 2021 Dec 1;116(12):2399-2409. doi: 10.14309/ajg.0000000000001375. PMID 34382947

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 112 subjects signed consent and randomized. Ten subjects screen failed prior to day 1 dosing ( after signing consent) and the number of participants who started the study is 102 subjects.
Period: Overall Study
Arm/Group | AXA1957 High Dose | AXA1957 Low Dose | AXA1125 | Placebo
Started | 32 | 26 | 29 | 15
Completed | 20 | 18 | 26 | 13
Not Completed | 12 | 8 | 3 | 2
Not completed — Adverse Event | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Subject noncompliance | 7 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is the safety analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | AXA1957 High Dose | AXA1957 Low Dose | AXA1125 | Placebo | Total
Number analyzed (Participants) | 32 | 26 | 29 | 15 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (12.79) | 49.6 (10.74) | 49.2 (12.79) | 53.2 (9.62) | 50.2 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 17 | 10 | 62
  Male | 13 | 10 | 12 | 5 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 1 | 5
  White | 31 | 24 | 26 | 14 | 95
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 26 | 29 | 15 | 102
Type 2 diabetes mellitus status (T2DM) [Count of Participants; unit: Participants] | 12 | 10 | 12 | 6 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Incidence of Study Product Emergent Adverse Events (AEs) and Any Serious Adverse Events (SAEs)
Description: Subjects received AXA1125 at 24 g twice daily ( BID), AXA1957 at 20.3 g BID or 13.5 g BID with Product related AEs and any SAEs up to 16 weeks
Time Frame: Baseline to week 16
Population: Subjects received AXA1125 at 24 g BID, AXA1957 at 20.3 g BID or 13.5 g BID, or placebo for up to 16 weeks.
Measure: Number; unit: participants
Arm/Group | AXA1957 High Dose | AXA1957 Low Dose | AXA1125 | Placebo
Number analyzed (Participants) | 32 | 26 | 29 | 15
participants
  Any Product Related Product-Emergent AEs | 10 | 8 | 13 | 2
  Any SAEs | 1 | 0 | 1 | 0

2. Secondary Outcome: Percent Change in Liver Fat as Assessed by MRI- Proton Density Fat Fraction (PDFF)
Description: Relative Changes From Baseline in MRI-PDFF at Week 16 in Overall Subjects (Safety Analysis Population)
Time Frame: Baseline to week 16
Population: Relative Changes From Baseline in MRI-PDFF at Week 16 in Overall Subjects (Safety Analysis Population)
Measure: Mean (Standard Deviation); unit: percentage of change of MRI_PDFF
Arm/Group | AXA1957 High Dose | AXA1957 Low Dose | AXA1125 | Placebo
Number analyzed (Participants) | 32 | 26 | 29 | 15
percentage of change of MRI_PDFF | -8.12 (24.904) | -20.29 (23.064) | -22.88 (23.040) | -5.74 (20.425)

3. Secondary Outcome: Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Description: Absolute Changes From Baseline in HOMA-IR at Week 16 in Overall Subjects (Safety Analysis Population)
Time Frame: Baseline to week 16
Population: Absolute Changes From Baseline in HOMA-IR at Week 16 in Overall Subjects (Safety Analysis Population)
Measure: Mean (Standard Deviation); unit: percentage of change of HOM-IR
Arm/Group | AXA1957 High Dose | AXA1957 Low Dose | AXA1125 | Placebo
Number analyzed (Participants) | 32 | 26 | 29 | 15
percentage of change of HOM-IR | 8.421 (34.5866) | 1.445 (3.6396) | -4.369 (16.8680) | 0.720 (4.7074)

4. Secondary Outcome: Change in Glucose Homeostasis
Description: Absolute Changes From Baseline in HbA1c at Week 16 in Subjects with Diabetes (Safety Analysis Population)
Time Frame: Baseline to week 16
Population: Absolute Changes From Baseline in HbA1c at Week 16 in Subjects with Diabetes (Safety Analysis Population)
Measure: Mean (Standard Deviation); unit: change in HbA1c
Arm/Group | AXA1957 High Dose | AXA1957 Low Dose | AXA1125 | Placebo
Number analyzed (Participants) | 9 | 9 | 11 | 3
change in HbA1c | 0.0138 (0.01419) | .0001 (0.00588) | -0.0070 (8.008) | -0.0027 (0.00874)

5. Secondary Outcome: Relative Change in Alanine Aminotransferase (ALT)
Description: Relative Changes From Baseline in ALT at Week 16 in Overall Subjects (Safety Analysis Population)
Time Frame: Baseline to week 16
Population: Relative Changes From Baseline in ALT at Week 16 in Overall Subjects (Safety Analysis Population)
Measure: Mean (Standard Deviation); unit: percentage change of ALT
Arm/Group | AXA1957 High Dose | AXA1957 Low Dose | AXA1125 | Placebo
Number analyzed (Participants) | 32 | 26 | 29 | 15
percentage change of ALT | -20.65 (30.163) | -19.19 (30.559) | -21.86 (25.991) | -7.20 (36.483)

6. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: Relative Changes From Baseline in AST at Week 16 in Overall Subjects (Safety Analysis Population)
Time Frame: Baseline to Week 16
Population: Relative Changes From Baseline in AST at Week 16 in Overall Subjects (Safety Analysis Population)
Measure: Mean (Standard Deviation); unit: percentage of AST from basline
Arm/Group | AXA1957 High Dose | AXA1957 Low Dose | AXA1125 | Placebo
Number analyzed (Participants) | 32 | 26 | 29 | 15
percentage of AST from basline | -13.40 (30.898) | -17.02 (30.898) | -16.76 (27.908) | -7.49 (40.499)

ADVERSE EVENTS:
Time Frame: From the time of informed consent up to first administration of study product on Day 1, any untoward medical occurrence considered related to study procedures will be recorded as an AE. Adverse events that occur from the first administration of study product on Day 1 through the Follow-up Visit / Week 18 will be considered treatment-emergent AEs
Arm/Group | AXA1957 High Dose | AXA1957 Low Dose | AXA1125 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/26 | 0/29 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/26 | 1/29 | 0/15
Other Adverse Events (participants affected / at risk) | 10/32 | 8/26 | 13/29 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXA1957 High Dose (N=32) | AXA1957 Low Dose (N=26) | AXA1125 (N=29) | Placebo (N=15)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AXA1957 High Dose (N=32) | AXA1957 Low Dose (N=26) | AXA1125 (N=29) | Placebo (N=15)
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 10 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 3 | 0
Headache (Nervous system disorders) | 2 | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04073368/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04073368/SAP_001.pdf